CLINICAL TRIAL: NCT02361320
Title: Imaging Biomarkers in Pancreatic and Hepatobiliary Cancers
Brief Title: Computed Tomography in Diagnosing Patients With Pancreatic or Hepatobiliary Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PA14-0319; NCI-2018-02642 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA14-0319 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-02-04; First posted 2015-02-11 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Pancreatic ductal adenocarcinoma; PDAC; Computed tomography; CT; Questionnaire; Survey
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Computed Tomography Scans (CT) (Experimental): Participants to receive 2 computed tomography (CT) scans that are part of their regular cancer care. One (1) scan performed before the start of chemotherapy, and the other at first restaging visit with oncologist. Participant to complete the MD Anderson Symptom Inventory for Gastrointestinal cancer (MDASI-GI) questionnaire at baseline visit, and follow up visit.
  Interventions: Procedure: Computed Tomography (CT); Behavioral: Questionnaire

INTERVENTIONS:
Procedure: Computed Tomography (CT) — Participants to receive 2 CT scans. One scan performed before the start of chemotherapy, and the other at first restaging visit with oncologist.
  Other Names: CT
Behavioral: Questionnaire — Participant to complete the MD Anderson Symptom Inventory for Gastrointestinal cancer (MDASI-GI) questionnaire at baseline visit, and follow up visit. Questionnaires should take about 10 minutes to complete.
  Other Names: Survey

SUMMARY:
This trial studies how well computed tomography works in diagnosing patients with pancreatic or hepatobiliary cancer. Computed tomography may help researchers predict how patients with pancreatic or hepatobiliary cancer may respond to chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To prospectively validate our pilot data that indicate that pre-therapy computed tomography-based (CT) mass transport properties correlate with overall survival.

II. To prospectively validate our pilot data that indicate that local control of pancreatic and hepatobiliary tumors correlate with changes in computed tomography-based mass transport properties of the tumors after cytotoxic therapies.

OUTLINE:

Patients undergo CT scan at baseline and after 4 to 6 cycles of fluorouracil/irinotecan/leucovorin calcium/oxaliplatin, or after 4 infusions of gemcitabine/nab-paclitaxel (or other gemcitabine-based regimens), or 6 to 12 weeks after radiotherapy for hepatobiliary cancers. Patients may undergo optional magnetic resonance imaging (MRI) scans prior to therapy, after two weeks of therapy, and at the time of the first restaging CT scan.

ELIGIBILITY:
Inclusion Criteria:

* PANCREATIC CANCER: Histologically confirmed adenocarcinoma of the pancreas
* PANCREATIC CANCER: Non-distant metastatic pancreatic cancer that is either

  * Unresectable locally advanced disease, defined as primary tumor that involves > 180 degrees of the superior mesenteric artery, celiac axis or any of its branches on CT or MRI, primary tumor that occludes the superior mesenteric vein or portal vein, aorta or inferior vena cava invasion, or superior mesenteric vein invasion below the transverse mesocolon
  * Borderline resectable disease, defined as primary tumor that involves =< 180 degrees of the superior mesenteric artery, celiac axis or any of its branches on CT or MRI, primary tumor that involves the superior mesenteric vein causing vein deformity or segmental venous occlusion with a patent vessel above and below suitable for reconstruction, or primary tumor that abuts or encases (>= 50% of the vessel circumference) a short segment of the common hepatic artery (typically at the gastroduodenal artery origin)
* PANCREATIC CANCER: Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1
* PANCREATIC CANCER: Women of childbearing potential (those who have not undergone a hysterectomy or who have not been postmenopausal for at least 24 consecutive months) must agree to practice adequate contraception and to refrain from breast feeding
* PANCREATIC CANCER: Patient who has been recommended chemotherapy treatment for pancreatic cancer
* PANCREATIC CANCER: Signed study-specific consent form
* HEPATOBILIARY CANCER: Diagnosis of

  * Hepatocellular carcinoma: This may be diagnosed in the following ways:

    * Pathologically (histologically or cytologically) proven diagnosis of hepatocellular carcinoma (HCC)
    * At least one solid liver lesion with arterial enhancement and washout on a delayed phase of a multi-phasic CT or MRI in the setting of cirrhosis or chronic hepatitis B or C without cirrhosis
  * Intrahepatic cholangiocarcinoma: Pathologically (histologically or cytologically) proven diagnosis of intrahepatic cholangiocarcinoma
* HEPATOBILIARY CANCER: Patients may have single or multinodular tumors
* HEPATOBILIARY CANCER: ECOG PS 0-1
* HEPATOBILIARY CANCER: Women of childbearing potential (those who have not undergone a hysterectomy or who have not been postmenopausal for at least 24 consecutive months) must agree to practice adequate contraception
* HEPATOBILIARY CANCER: Prior history of surgical resection, chemotherapy, transarterial chemoembolization (TACE), and/or radiofrequency ablation are allowed
* HEPATOBILIARY CANCER: Patients may be enrolled if:

  * The patient is dispositioned to receive definitive radiotherapy
  * The patient has received definitive radiotherapy within the past two years and has liver protocol CT or MRI scans before radiotherapy and at first restaging after radiotherapy
* HEPATOBILIARY CANCER: Signed study-specific consent form

Exclusion Criteria:

* Presence of distant metastasis
* Patients whose tumors are defined as resectable
* Unstable angina or New York Heart Association grade II or greater congestive heart failure
* Evidence of fever or acute infection (chronic infection such as hepatitis virus is acceptable)
* Coexisting medical condition that would preclude chemotherapy, radiotherapy, or iodine-based contrast enhanced CT scan
* Pregnant women with a positive pregnancy test
* Inability to comply with study and/or follow-up procedures
* Patients with an active second malignancy with the exception of non-melanoma skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Estimated)
Dates: Start 2015-03-09 (Actual); Primary Completion 2026-06-27 (Estimated); Study Completion 2026-06-27 (Estimated)

PRIMARY OUTCOMES:
Correlation Between Local Control and Changes in Mass Transport by Computed Tomography (CT) | 4 months
  Local tumor progression defined by clinical signs or symptoms of local pancreatic tumor growth (e.g., worsening back/abdominal pain, obstruction, jaundice, etc.) that are documented by the attending clinician and research data coordinator and/or diagnostic imaging evidence of tumor growth. Kaplan-Meier method used to estimate probabilities of LPFS for patients with a normalized AUC ratio <1 and patients with a normalized AUC ratio >/=1, respectively. Log rank test applied to compare the LPFS between these two patient groups. Multivariate Cox proportional hazards models fitted to compare the LPFS between the two comparison groups, adjusting for the effects of patients' characteristics and clinical factors.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Koay, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org